CLINICAL TRIAL: NCT01499797
Title: Towards a CARE AND WELFARE STANDARD for Community-dwelling Frail Elderly People With Complex Health Problems
Brief Title: The CareWell-programme for Community-dwelling Frail Elderly Persons.
Acronym: CareWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Healthcare Authority (Unknown); Health insurances CZ (Unknown); Health insurances UVIT (Unknown); City of Nijmegen (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010/403
Record Dates: First submitted 2011-10-20; First posted 2011-12-26 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2011-10

CONDITIONS: Overall Functioning; Incremental Cost-effectiveness Ratio
Keywords: frailty; frail elders; multicomponent intervention; overall functioning; cost-effectiveness; integrated care; primary care; community dwelling
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- regular medical care (No Intervention): Identified community dwelling frail elderly people receiving regular medical care in their primary care setting
- The CareWell programme (Experimental): Identified community dwelling frail elderly people receiving care in line with the CareWell programme
  Interventions: Other: The CareWell programme

INTERVENTIONS:
Other: The CareWell programme — The CareWell programme contains the following components:
  * multidisciplinary primary care teams
  * working with proactive care plans integrating cure, care and welfare
  * advanced care planning (e.g. recording limitations of treatment, non-resuscitation decisions)
  * medication review
  * case-management
  * guidelines for consultation of in-hospital geriatric experts
  * guidelines for transfers from primary care to home-based facilities and hospital and back
  * practice guidelines for management of common geriatric conditions
  Other Names: Multi-component intervention for frail elderly; Integrated care for community-dwelling frail elderly
  Arms: The CareWell programme

SUMMARY:
The purpose of this study is to investigate the effect of the CareWell-programme on overall functioning of community-dwelling frail elderly persons. Furthermore, the total costs and the cost-effectiveness of the CareWell-programme, in comparison with regular medical care, will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Frail community dwelling elderly patients aged 70 years or above. Frailty is determined with a two-phase screening instrument.

Exclusion Criteria:

* Non-frail elders
* Patients in palliative or end-of-life stages of disease
* Patients residing in long-term care facilities (care homes and nursing homes)
* Patients already enrolled in specific dementia-related case-management programmes who lack other health-related problems
* Patients not speaking or understanding the Dutch language

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 536 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Overall functioning | 18 months
  Overall functioning is measured with the Katz-15 questionnaire. Katz-15 is embedded in the minimal data set (MDS). This MDS is used by all research projects of the Dutch National Program on Elderly Care
Incremental cost-effectiveness ratio (ICER) | 18 months

SECONDARY OUTCOMES:
Perceived quality of life | 18 months
  Perceived quality of life is measured with the RAND-36 questionnaire. RAND-36 is embedded in the minimal data set (MDS). This MDS is used by all research projects of the Dutch National Program on Elderly Care
Psychological well-being | 18 months
  Psychological well-being is measured with the RAND-36 questionnaire.
Social functioning | 18 months
  Social functioning is measured with the RAND-36 questionnaire.
Perceived health | 18 months
  Perceived health is measured with the RAND-36 questionnaire abd Cantril's Self Anchoring Ladder. Both RAND-36 as Cantril's Self Anchoring Ladder are embedded in the minimal data set (MDS).
Utility | 18 months
  Utility is measured with the EQ-5D questionnaire. EQ-5D is embedded in the minimal data set (MDS).
Health care consumption | 18 months
  Health care consumption including hospital resource consumption, unplanned GP care (evenings, nights and weekends), home care, temporary or permanent admission to a residential care home, temporary or permanent admission to a nursing home, day care, visits to outpatients'clinics.
Use of welfare services | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Koopmans, Professor, Principal Investigator — Radboud University Medical Center
Locations (10):
- Netherlands (10):
  - Huisartsengroep Milbergen (van der Ligt/ Krijgsman), Oude Gracht 16, Beek-Ubbergen
  - Gezondheidscentrum de Kroonsteen, Schoolstraat 8, Malden
  - Gezondheidscentrum de Vuursteen, Prinsenweg 6, Molenhoek
  - Medisch Centrum Brakkenstein, Kanunnik Boenenstraat 8, Nijmegen
  - Gezondheidscentrum Hazenkamp, Vossenlaan 76, Nijmegen
  - Huisartsenpraktijk Jacobslaan (Dreijerink/ van der Laan-Evers), Jacobslaan 345, Nijmegen
  - Huisartsenpraktijk de Haterse HOED, Couwenbergstraat 34-36, Nijmegen
  - Huisartsenpraktijk Danielsplein, Danielsplein 4, Nijmegen
  - Medipark (Graat), Hyacinthstraat 3a, Uden
  - Huisartsenpraktijk Ubachs/Vogels, Huissteden 1450, Wijchen

REFERENCES:
- [Derived] Ruikes FGH, Adang EM, Assendelft WJJ, Schers HJ, Koopmans RTCM, Zuidema SU. Cost-effectiveness of a multicomponent primary care program targeting frail elderly people. BMC Fam Pract. 2018 May 16;19(1):62. doi: 10.1186/s12875-018-0735-4. PMID 29769026
- [Derived] Ruikes FG, Meys AR, van de Wetering G, Akkermans RP, van Gaal BG, Zuidema SU, Schers HJ, van Achterberg T, Koopmans RT. The CareWell-primary care program: design of a cluster controlled trial and process evaluation of a complex intervention targeting community-dwelling frail elderly. BMC Fam Pract. 2012 Dec 5;13:115. doi: 10.1186/1471-2296-13-115. PMID 23216685